CLINICAL TRIAL: NCT03940235
Title: Radioablation +/- Hormonotherapy for Prostate Cancer Oligorecurrences (RADIOSA Trial): Potential of Imaging and Biology
Brief Title: Radioablation With or Without Androgen DeprIvation Therapy in Metachronous Prostate Cancer OligometaStAsis
Acronym: RADIOSA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO 997
Record Dates: First submitted 2019-04-24; First posted 2019-05-07 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Oligometastatic Prostate Cancer
MeSH Terms: interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic body Radiotherapy (SBRT) only (Experimental): ARM 1: salvage SBRT for lymph nodes and/or bone metastases. All the radiologically documented lesions will be treated simultaneously.
  Interventions: Radiation: SBRT
- Stereotactic body Radiotherapy (SBRT) and hormonotherapy (ADT) (Active Comparator): ARM 2: salvage SBRT (as described for ARM 1) + 6-month ADT (luteinizing hormone-releasing hormone (LHRH) agonist or antagonist). ADT should start within one week before the start of SBRT.
  Interventions: Drug: Androgen deprivation therapy (ADT); Radiation: SBRT

INTERVENTIONS:
Drug: Androgen deprivation therapy (ADT) — SBRT + ADT
  Arms: Stereotactic body Radiotherapy (SBRT) and hormonotherapy (ADT)
Radiation: SBRT — SBRT to all radiological documented lesions (bone or lymphnodes)

SUMMARY:
A randomized phase II clinical trial (RADIOSA trial: Radioablation with or without Androgen DeprIvation therapy in metachronous prostate cancer OligometaStAsis).

The aim is to compare time to progression between the two study arms: SBRT only or SBRT and hormonotherapy (ADT). The primary objective is to compare the progression-free survival (PFS) defined as the absence of new metastatic lesions (local, regional or distant) between the two arms. The secondary endpoints include the comparison of overall survival (OS), biochemical progression-free survival (BPFS), ADT-free survival, local control, treatment-induced acute and late toxicity, time to castration-resistant disease and QoL between the two arms; the development of a dedicated biobanking (collection of plasma and serum) for further biological investigation of predictive/diagnostic factors for personalized treatment; the preliminary evaluation of prognostic biomarkers; the correlation between imaging-derived parameters and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of adenocarcinoma of the prostate;
* Biochemical relapse of PCa following radical local prostate treatment (radical prostatectomy, primary radiotherapy or radical prostatectomy +/- prostate bed adjuvant/salvage radiotherapy) +/- ADT according to the European Association of Urology (EAU) guidelines 2016 [18] or after any salvage therapy if biochemical progression is diagnosed in the context of castration sensitive PCa;
* Nodal relapse in the pelvis, extra-regional nodal relapse (M1a), bone metastases (M1b) on Ch-PET/CT or WBMRI with a maximum of 3 lesions;
* Serum testosterone level >50 ng/dl at the time of randomization (castration sensitive PCa)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Age ≥18 years;
* Written informed consent signed

Exclusion criteria

* Serious concomitant comorbidities or contraindication to SBRT and/or ADT;
* Previous invasive cancer (within 3 years before the prostate cancer diagnosis) apart from non-melanoma skin malignancies;
* No ability to complete questionnaires about QoL;
* Presence of mental diseases that cannot ensure valid informed consent;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up 3 months from the end of the treatment up to radiological progression within 3 years
  Defined as the absence of new metastatic lesions (local, regional or distant) between the two arms.

SECONDARY OUTCOMES:
Overall survival (OS) | Up the end of SBRT until death for cancer or other causes up to 3 years
  From the end of RT treatment to the time of clinical progression or mortality from specific disease cause
Biochemical progression-free survival (BPFS) | up 3 months from the end of the treatment up to 3 years
  Biochemical progression is defined according to the EAU guidelines [18], namely a rising PSA level >0.2 ng/ml following radical prostatectomy and >2 ng/ml above the nadir after radiation therapy.
Numbers of patients who experienced acute and late toxicity | Up to 1 months after treatment completion and then up to 3 years
  Toxicity will be assessed according to the Common Toxicity Criteria for adverse events (CTCAE) toxicity criteria v4.3

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Jereczek-Fossa, Prof, Study Director — Istituto Europeo di Oncologia IRCCS Milan, Italy
Locations (1):
- Istituto Europeo di Oncologia IRCCS, Milan, MI - Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vavassori A, Mauri G, Mazzola GC, Mastroleo F, Bonomo G, Durante S, Zerini D, Marvaso G, Corrao G, Ferrari ED, Rondi E, Vigorito S, Cattani F, Orsi F, Jereczek-Fossa BA. Cyberknife Radiosurgery for Prostate Cancer after Abdominoperineal Resection (CYRANO): The Combined Computer Tomography and Electromagnetic Navigation Guided Transperineal Fiducial Markers Implantation Technique. Curr Oncol. 2023 Aug 28;30(9):7926-7935. doi: 10.3390/curroncol30090576. PMID 37754491
- [Derived] Carloni G, Garibaldi C, Marvaso G, Volpe S, Zaffaroni M, Pepa M, Isaksson LJ, Colombo F, Durante S, Lo Presti G, Raimondi S, Spaggiari L, de Marinis F, Piperno G, Vigorito S, Gandini S, Cremonesi M, Positano V, Jereczek-Fossa BA. Brain metastases from NSCLC treated with stereotactic radiotherapy: prediction mismatch between two different radiomic platforms. Radiother Oncol. 2023 Jan;178:109424. doi: 10.1016/j.radonc.2022.11.013. Epub 2022 Nov 24. PMID 36435336
- [Derived] Marvaso G, Ciardo D, Corrao G, Gandini S, Fodor C, Zerini D, Rojas DP, Augugliaro M, Bonizzi G, Pece S, Cattani F, Mazzocco K, Mistretta FA, Musi G, Alessi S, Petralia G, Pravettoni G, De Cobelli O, Di Fiore PP, Viale G, Orecchia R, Jereczek-Fossa BA. Radioablation +/- hormonotherapy for prostate cancer oligorecurrences (Radiosa trial): potential of imaging and biology (AIRC IG-22159). BMC Cancer. 2019 Sep 10;19(1):903. doi: 10.1186/s12885-019-6117-z. PMID 31500605